CLINICAL TRIAL: NCT06510101
Title: Manual Manipulation and Ex Vivo Flexible Ureteroscopic Lithotripsy to Salvage Deceased Donor Kidneys With Renal Stones: A Case Series
Status: Enrolling by invitation | Type: Observational
Sponsor: Yingxin FU.MD (Other)
Collaborators: Shenzhen Third People's Hospital (Other); The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor-Investigator, Yingxin FU.MD, Head of department, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Other Study IDs: MMEVFUL
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Manual Manipulation and Ex Vivo Flexible Ureteroscopic Lithotripsy to Salvage Deceased Donor Kidneys With Renal Stones:a New Method by
Keywords: organ donation;; kidney transplantation; flexible ureteroscopy;

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
we report the manual manipulation and Ex Vivo Flexible Ureteroscopic Lithotripsy to Salvage Deceased Donor Kidneys with Renal Stones,including nine cases,Renal transplantation was performed with the treated kidney after removing the stones, and the short-term postoperative outcomes were promising. cases were thoroughly reported in this paper.

DETAILED DESCRIPTION:
The presence of donor kidney stones may lead to ureteral obstruction after transplantation, affecting the recovery of postoperative renal function. Thus, donors with kidney stones are often considered marginal kidney donors and likely disqualified,Here we describe a series case of multiple kidney stones in a donor kidney treated with the combined application of fURS and holmium laser lithotripsy (HLL) before transplantation. Renal transplantation was performed with the treated kidney after removing the stones, and the short-term postoperative outcomes were promising. The case was thoroughly reported in this paper.

ELIGIBILITY:
Inclusion Criteria:

* get renal transplantation donor kidney with stones

Exclusion Criteria:

* without renal stones the renal stones without Ex Vivo Flexible Ureteroscopic Lithotripsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patinet in our centor get a ranal transplantation with stones
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
eGFR | 3monthes after transplantation
  renal function

CONTACTS AND LOCATIONS:
Locations (1):
- yingxin Fu, Shenzhen, Guangdong, China